CLINICAL TRIAL: NCT04232163
Title: Evaluation of a Program to Increase Upper Limb Recovery After Stroke
Brief Title: Arm Boot Camp Study: Evaluation of a Program to Increase Upper Limb Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H19-02005
Record Dates: First submitted 2019-12-23; First posted 2020-01-18 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Ischemia; Brain Infarction; Vascular Diseases; Infarction; Nervous System Diseases; Cardiovascular Diseases
Keywords: Stroke; Upper extremity; Rehabilitation; Wearable device; Exercise; Randomized Controlled Trial
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Ischemia; Brain Infarction; Vascular Diseases; Infarction; Nervous System Diseases; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): Participants will receive the intervention right away
  Interventions: Behavioral: Arm Boot Camp
- Delayed Treatment Group (No Intervention): Participants will receive usual care (no intervention), however, they will receive the intervention after a 3 week delay

INTERVENTIONS:
Behavioral: Arm Boot Camp — The intervention involves a combination of daily homework based upper limb exercises and feedback from an activity monitor to motivate use of the affected upper limb. Participants will be supported through virtual sessions with a therapist.
  Arms: Immediate Treatment Group

SUMMARY:
This study will examine the feasibility and effect of a program that combines exercise and feedback from a wearable device on upper limb movement practice and function in individuals with stroke.

DETAILED DESCRIPTION:
Participants will be randomized into either the Immediate Treatment Group or the Delayed Treatment group. Both groups will complete the same intervention program. The Immediate treatment group will start the program right away while the Delayed Treatment group will start the program after a 3 week delay. The intervention program is 3 weeks in duration and consists of participants completing at least two hours of exercises (adapted from the Home-GRASP program) daily and wearing an activity monitor on their affected wrist during waking hours for the duration of the intervention. Participants will be asked to meet daily movement count goals based on information from the monitor. Participants will have 6 virtual sessions with a therapist who will teach and monitor exercises thru an online platform (Zoom Video Communications), work with participants to generate and progress daily movement goals and discuss barriers and potential solutions to exercise adherence and/or meeting movement goals.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* < 1 year since the stroke occurred
* Living in the community
* Have unilateral upper limb impairment
* Have some ability to move their arm and hand (> 30° shoulder flexion or abduction and Fugl Meyer finger extension score > 0)
* Are using their affected upper limb in a different way than prior to their stroke (REACH score < 4)
* Completed formal physical and occupational therapy rehabilitation for the upper limb
* Have access to a tablet, computer, laptop or phone with internet and email access.

NOTE: If participant have a caregiver, we would like to invite him/her to assist in this study; however, a caregiver is not a must for participating in this study.

Exclusion Criteria:

* musculoskeletal/other neurological conditions that limit movement in their arm
* unable to provide informed consent
* have another medical condition that would affect their ability to participate in the treatment protocol
* have persistent pain in their affected upper limb that affects their ability to use the limb
* Unable to speak, understand, or read English (unless another person, [i.e., family member, care taker or friend] can be present and translate during measurement/treatment sessions, and home activities related to the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Hand counts captured using an activity monitor | Post intervention (immediately following 3 weeks of intervention)
  Participants wear the activity monitor on stroke affected arm during waking hours for 3 consecutive days

SECONDARY OUTCOMES:
ArmCAM (Arm Capacity and Movement Test) | Post intervention (immediately following 3 weeks of intervention), follow up (2 months after completion of intervention)
  The online upper extremity functional assessment consists of 10 items that measure gross movements, supported reach, functional reach and grasp movements, functional wrist movement, and fine motor skills.
Stroke Impact Scale - hand and strength scales | Post intervention (immediately following 3 weeks of intervention), follow up (2 months after completion of intervention)
  Evaluate how stroke has impacted health and life
Hand count measured during the intervention sessions | Daily counts within 3 week intervention
  Daily hand count data captured using activity monitor on the stroke affected arm during intervention period
REACH Scale | Post intervention (immediately following 3 weeks of intervention), follow up (2 months after completion of intervention)
  A self-report measure for individuals with stroke that captures how the affected arm and hand is being used outside of the clinical setting.
Hand counts captured using an activity monitor | Follow up (two months after completion of intervention)
  Participants wear the activity monitor on stroke affected arm during waking hours for 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, PhD, Principal Investigator — University of British Columbia
Locations (7):
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - GF Strong Rehab Centre, Vancouver, British Columbia
  - Riverview Health Centre, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson LA, Mow A, Menon C, Eng JJ. Preliminary Examination of the Ability of a New Wearable Device to Capture Functional Hand Activity After Stroke. Stroke. 2019 Dec;50(12):3643-3646. doi: 10.1161/STROKEAHA.119.026921. Epub 2019 Oct 30. PMID 31662119
- [Derived] Simpson LA, Barclay R, Bayley MT, Brasher PMA, Dukelow SP, MacIntosh BJ, MacKay-Lyons M, Menon C, Mortenson WB, Peng TH, Pollock CL, Pooyania S, Silverberg ND, Teasell R, Yao J, Eng JJ. A Randomized Control Trial of a Virtually Delivered Program for Increasing Upper Limb Activity After Stroke. Neurorehabil Neural Repair. 2025 Mar;39(3):179-189. doi: 10.1177/15459683241303702. Epub 2024 Dec 27. PMID 39727287
- [Derived] Simpson LA, Barclay R, Bayley MT, Dukelow SP, MacIntosh BJ, MacKay-Lyons M, Menon C, Mortenson WB, Peng TH, Pollock CL, Pooyania S, Teasell R, Yang CL, Yao J, Eng JJ. Virtual Arm Boot Camp (V-ABC): study protocol for a mixed-methods study to increase upper limb recovery after stroke with an intensive program coupled with a grasp count device. Trials. 2022 Feb 8;23(1):129. doi: 10.1186/s13063-022-06047-9. PMID 35135585